CLINICAL TRIAL: NCT06144918
Title: A Phase 2, Double-Masked, Randomized, Placebo-Controlled, Dose-Response Study Assessing the Safety and Ocular Hypotensive Efficacy of Two Concentrations of SBI-100 Ophthalmic Emulsion in Patients With Elevated Intraocular Pressure
Brief Title: Ph2 Placebo-Controlled Study for Safety & Ocular Efficacy of SBI-100 Ophthalmic Emulsion in Pts w/ Elevated Eye Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Skye Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBI-100-201
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Results first posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-05

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: glaucoma; IOP; ocular hypertension; POAG
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SBI-100 Ophthalmic Emulsion, 0.5% (Experimental): All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 Ophthalmic Emulsion
  Interventions: Drug: SBI-100 Ophthalmic Emulsion, 0.5%
- SBI-100 Ophthalmic Emulsion Placebo (Placebo Comparator): All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 Ophthalmic Emulsion
  Interventions: Drug: SBI-100 Ophthalmic Emulsion, Placebo
- SBI-100 Ophthalmic Emulsion, 1% (Experimental): All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 Ophthalmic Emulsion
  Interventions: Drug: SBI-100 Ophthalmic Emulsion, 1.0%

INTERVENTIONS:
Drug: SBI-100 Ophthalmic Emulsion, 0.5% — 0.5% (5 mg/mL) SBI-100 Ophthalmic Emulsion eyedrop
  Arms: SBI-100 Ophthalmic Emulsion, 0.5%
Drug: SBI-100 Ophthalmic Emulsion, 1.0% — 1.0% (10 mg/mL) SBI-100 Ophthalmic Emulsion eyedrop
  Arms: SBI-100 Ophthalmic Emulsion, 1%
Drug: SBI-100 Ophthalmic Emulsion, Placebo — Placebo, SBI-100 Ophthalmic Emulsion eyedrop without the active ingredient (SBI-100)
  Arms: SBI-100 Ophthalmic Emulsion Placebo

SUMMARY:
The goal of this clinical trial is to test in patients with glaucoma and elevated pressure in the eye. The main questions it aims to answer are: • ability to lower pressure in the eye • safety in the eye and the body of patients with elevated pressure in the eye. Patients will be randomly given either:

* 0.5% (5 mg/mL) SBI-100 Ophthalmic Emulsion
* 1.0% (10 mg/mL) SBI-100 Ophthalmic Emulsion
* Placebo Ophthalmic Emulsion

Patients will be tested before starting and will have one drop of the product placed into each eye twice a day for 14 days, by the site and by the patient. At the end of the study, researchers will compare the groups to see if there is a change from before use of SBI-100 Ophthalmic Emulsion to the end of study.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-masked, placebo-controlled Phase 2 study to evaluate the ocular hypotensive efficacy, safety, and tolerability of SBI-100 Ophthalmic Emulsion after 14 days of binocular dosing, twice daily (BID).

There will be a 35-day screening period, including wash-out (if needed), followed by a visit on Day-1 to confirm eligibility. The first dose will be administered by the staff immediately after the (eligibility) 08:00 IOP measurement on Day 1, with subsequent study assessments up to 8 hours post-dose. The PM (evening) dose will be self-administered by the patient at home, approximately 12 hours after the AM (morning) dose. The patient will self-administer study treatment on Days 2 through 6 in the AM and PM. On Day 7, the patient will return to have the AM dose administered by site staff immediately after the 08:00 IOP measurement has been taken. Subsequent assessments will be performed in a similar fashion as Day 1 with study assessments up to 8 hours post-dose. Patient will self-administer the Day 7 PM dose and the AM and PM doses on Days 8 through 13. On Day 14, the patient will return to have the AM dose administered by site and assessments similar to that of Days 1 and 7, the patient may complete the final dose on Day 14 at the site approximately 12 hours after the AM dose and have end of study (EOS) procedures performed. Or the patient may choose to self-administer the Day 14 PM dose at home and return to the site within 2 days for EOS visit.IOP efficacy will be evaluated by Goldmann applanation tonometry. Safety/tolerability will be evaluated by review of ocular signs and symptoms through Best Corrected Visual Acuity (BCVA), ophthalmic assessments, ocular comfort patient-reported outcome (PRO), vital signs, and other standard safety measures

Diagnosis and main criteria for inclusion: Patients with primary open-angle glaucoma (POAG) or ocular hypertension (OHT)

Screening: up to 35 days, including wash-out from any topical pharmacological IOP-lowering therapies (if required) Treatment: 2 weeks (14 days) Follow up: Up to 2 days after the last dose on Day 14

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age or greater at time of informed consent.
2. Diagnosis of either primary open angle glaucoma (POAG) or ocular hypertension (OHT) in each eye.
3. Intraocular Pressure (IOP) Criteria:

   1. If currently on an IOP-lowering therapy, patient is willing to withhold therapy according to study requirements, and in the opinion of the Investigator, can do so without significant risk.
   2. If treatment naïve, Screening IOP is ≥ 21 and ≤ 36 mmHg in each eye, and in the opinion of the Investigator, is likely to be controlled on a single IOP-lowering therapy.
   3. 08:00 Hour IOP is between 21 and 36 mmHg in each eye on Day-1 and Day 1.
4. Central corneal thickness between 480 and 620 μm at Screening in each eye.
5. Best correct visual acuity (BCVA) for distance equivalent to 20/100 or better in each eye at Screening and Day 1 (pre-dose).

Exclusion Criteria:

Either eye:

1. Mean/Median intraocular pressure > 36 mmHg at Screening and/or any time prior to treatment administration.
2. Concurrent treatment for glaucoma requiring more than 2 topical therapies (either as 2 independent monotherapies or as fixed dose combination), oral IOP-lowering therapy and/or in the opinion of the Investigator cannot be controlled on a single IOP therapy.
3. Has planned ocular surgeries/procedures within the duration of the study.
4. Any occurrences of the following prior to Day 1:

   1. Ocular trauma or surgery within 6 months
   2. Ocular laser treatments within 3 months
   3. In the opinion of the Investigator history or evidence of clinically significant ocular inflammation, including but not limited to blepharitis, conjunctivitis, etc.
   4. History of recurrent ocular herpes (simplex or zoster)
   5. Previous glaucoma intraocular surgery or glaucoma laser procedure and/or refractive surgery (e.g., radial keratotomy, PRK, SLT, LASIK, etc.) within 6 months
   6. Ocular medication within 30 days prior, except for:

   i. IOP-lowering therapies (washed-out per study requirements) ii. Lid scrubs iii. Artificial tears, gels and/or ointments to treat dry eye disease that in the opinion of the Investigator is not considered chronic use
5. Visual field loss, in the opinion of the Investigator, is functionally significant
6. Will require contact lenses and cannot refrain from using them at least 7 days prior to Day 1 and throughout the study.

General/Systemic:

1. Participation in any investigational study within 30 days of screening.
2. Known hypersensitivity or allergic reaction to cannabinoids, cannabis, sesame seed/oil or any component of the SBI-100 Ophthalmic Emulsion formulation and/or topical anesthetics.
3. Females of childbearing potential (not confirmed as post-menopausal or surgically sterile within the 6 months prior to screening) who are pregnant, nursing, or planning a pregnancy during the study and not using a reliable method of contraception from screening until at least 30 days after the last dose.
4. Males with partners of childbearing potential and do not agree to use a reliable method of contraception during the study and at least 30 days after the last dose.
5. Patients with a history of substance or alcohol abuse, considered chronic tetrahydrocannabinol (THC) users and/or test positive for alcohol or illicit drug use at Screening or Day-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2023-11-09 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tu Diep, Study Chair — Skye Bioscience, Inc.
Locations (3):
- United States (3):
  - Global Research Management, Inc., Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a screening/washout period of up to 35 days to washout procedures and medications prohibited by the study protocol. At Visit 3 (Day 1), eligible patients were randomized 1:1:1 to IP in a double-masked fashion (SBI-100 0.5%, SBI-100 1.0% or placebo).
  Eleven (11) participants were screen failures and therefore, did not receive a treatment assigned. A total of 56 participants were screened and enrolled.
Units Other Than Participants: Eyes
Groups:
- SBI-100 Ophthalmic Emulsion, 0.5%: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 ophthalmic emulsion
  SBI-100 ophthalmic emulsion, 0.5%: 0.5% (5 mg/ml) SBI-100 ophthalmic emulsion
- SBI-100 Ophthalmic Emulsion 1.0%: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 ophthalmic emulsion
  SBI-100 ophthalmic emulsion, 1.0%: 1.0% (10 mg/ml) SBI-100 ophthalmic emulsion
- Placebo: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 ophthalmic emulsion
  Placebo
Period: Overall Study
Arm/Group | SBI-100 Ophthalmic Emulsion, 0.5% | SBI-100 Ophthalmic Emulsion 1.0% | Placebo
Started | 19; 19 Eyes | 19; 19 Eyes | 18; 18 Eyes
Completed | 19; 19 Eyes | 19; 19 Eyes | 18; 18 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SBI-100 Ophthalmic Emulsion, 0.5% | SBI-100 Ophthalmic Emulsion 1.0% | Placebo | Total
Number analyzed (Participants) | 19 | 19 | 18 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 4 | 14
  >=65 years | 12 | 16 | 14 | 42
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 11 | 28
  Male | 9 | 12 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 5 | 16
  Not Hispanic or Latino | 15 | 12 | 13 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 2
  White | 17 | 17 | 18 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 18 | 56
Diagnosis for Study Inclusion [Count of Participants; unit: Participants]
  OHT (ocular hypertension) | 9 | 4 | 9 | 22
  POAG (primary open angle glaucoma) | 7 | 15 | 8 | 30
  Both OHT and POAG | 3 | 0 | 1 | 4
Study Eye [Count of Participants; unit: Participants]
  OD (oculus dexter; right eye) | 10 | 11 | 13 | 34
  OS (oculus sinister; left eye) | 9 | 8 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Hypertension as Measured by Intraocular Pressure (IOP)
Description: To evaluate the diurnal ocular hypotensive efficacy of 2 dose levels of SBI-100 Ophthalmic Emulsion compared to placebo in patients with elevated Intraocular Pressure (IOP). IOP was measured by Goldmann applanation tonometry and values were compared between baseline and Day 14 (evaluation of mean change in mmHg (millimeters of mercury)).
Time Frame: baseline and day 14
Measure: Least Squares Mean (Standard Error); unit: Change in IOP mmHg
Groups:
- SBI-100 Ophthalmic Emulsion 1.0%: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% of placebo, SBI-100 ophthalmic emulsion.
  SBI-100 ophthalmic emulsion, 1.0%. 1.0% (10 mg/ml) SBI-100 ophthalmic emulsion
- Placebo: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% of placebo, SBI-100 ophthalmic emulsion.
  Placebo
Arm/Group | SBI-100 Ophthalmic Emulsion, 0.5% | SBI-100 Ophthalmic Emulsion 1.0% | Placebo
Number analyzed (Participants) | 19 | 19 | 18
Change in IOP mmHg | -1.985 (0.5039) | -1.118 (0.5041) | -0.827 (0.5177)

2. Primary Outcome: Ocular and Systemic Safety as Assessed by Treatment Emergent Adverse Events (TEAEs)
Description: To evaluate the ocular and systemic safety of SBI-100 Ophthalmic Emulsion in patients with elevated IOP. Safety and tolerability were evaluated by review of ocular signs and symptoms through use of BCVA (best corrected visual acuity; change in score from baseline to Day 14), ophthalmic assessments) including slit lamp biomicroscopy, dilated fundus exam, pupil diameter, visual field and pachymetry), ocular comfort patient reported outcome, vital signs, assessment of adverse events (ocular and non-ocular).
Time Frame: baseline up to day 16
Measure: Number; unit: Events
Groups:
- SBI-100 Ophthalmic Emulsion Placebo: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or placebo, SBI-100 ophthalmic emulsion. SBI-100 ophthalmic emulsion, Placebo: Placebo, SBI-100 ophthalmic emulsion eyedrop without the active ingredient (SBI-100)
- SBI-100 Ophthalmic Emulsion, 0.5%: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% of placebo, SBI-100 ophthalmic emulsion.
  SBI-100 ophthalmic emulsion, 0.5%: 0.5% (5 mg/ml) SBI-100 ophthalmic emulsion.
- SBI-100 Ophthalmic Emulsion 1.0%: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% of placebo, SBI-100 ophthalmic emulsion.
  SBI-100 ophthalmic emulsion, 1.0%: 1.0% (10 mg/ml) SBI-100 ophthalmic emulsion.
Arm/Group | SBI-100 Ophthalmic Emulsion Placebo | SBI-100 Ophthalmic Emulsion, 0.5% | SBI-100 Ophthalmic Emulsion 1.0%
Number analyzed (Participants) | 18 | 19 | 19
Events | 3 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline through end of study (approximately 16 days post first dose).
Groups:
- SBI-100 Ophthalmic Emulsion, 1.0%: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 ophthalmic emulsion
  SBI-100 ophthalmic emulsion, 1.0%: 1.0% (10 mg/ml) SBI-100 ophthalmic emulsion
- Placebo: All patients enrolled into the study will be randomly assigned to an interventional treatment of 0.5% or 1.0% or Placebo, SBI-100 ophthalmic emulsion
Arm/Group | SBI-100 Ophthalmic Emulsion, 0.5% | SBI-100 Ophthalmic Emulsion, 1.0% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 14/19 | 19/19 | 8/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBI-100 Ophthalmic Emulsion, 0.5% (N=19) | SBI-100 Ophthalmic Emulsion, 1.0% (N=19) | Placebo (N=18)
Bruised right hip secondary to fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye worsening (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Infections / nasopharyngitis / common cold (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Instillation site erythema / redness less than 1 minute (General disorders) | 1 (1) | 0 (0) | 0 (0)
Instillation site irritation / burning upon administration (General disorders) | 2 (2) | 3 (3) | 1 (1)
Instillation site irritation / burning less than one minute (General disorders) | 3 (3) | 6 (6) | 2 (2)
Instillation site irritation / burning for 15 minutes (General disorders) | 0 (0) | 1 (1) | 0 (0)
Instillation site irritation / burning up to 15 seconds (General disorders) | 0 (0) | 0 (0) | 1 (1)
Instillation site irritation / burning up to 5 minutes (General disorders) | 1 (1) | 0 (0) | 0 (0)
Instillation site irritation / stinging up on administration (General disorders) | 4 (4) | 5 (5) | 1 (1)
Instillation site irritation / stinging for 20 seconds (General disorders) | 4 (4) | 5 (5) | 1 (1)
Minor concussion secondary to fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ocular irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma right side face (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Subconjunctival hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vivid dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol (2023-09-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT06144918/Prot_001.pdf
  • Statistical Analysis Plan: Original, version 1.0 (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/18/NCT06144918/SAP_002.pdf
  • Statistical Analysis Plan: Version 2.0 (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT06144918/SAP_003.pdf
  • Informed Consent Form (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT06144918/ICF_004.pdf